CLINICAL TRIAL: NCT05214417
Title: Conscious Dying/Conscious Living: Ketamine-Assisted Psychotherapy (KAP) for Patients at End of Life-A Pilot Study for Palliative and Hospice Care
Brief Title: Conscious Dying/Conscious Living: Ketamine-Assisted Psychotherapy
Acronym: KRF-EOL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Ketamine Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRF-EOL
Record Dates: First submitted 2022-01-17; First posted 2022-01-28 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Illness Terminal
Keywords: ketamine; ketamine assisted psychotherapy; palliative care; hospice; death and dying; conscious dying; psychedelic psychotherapy; psychedelics; end of life; life threatening illnesses
MeSH Terms: conditions — Death

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KAP (Ketamine-assisted Psychotherapy) Recipients (Experimental): Two separate IM ketamine injection sessions, with possible multiple doses administered at each session not to exceed 100 mg IM ketamine total for the session.
  Interventions: Drug: Ketamine Injectable Solution
- Naturalistic Comparator (Other): Pre-existing conventional treatment will continue for this group during the study period.
  Interventions: Other: Naturalistic Control

INTERVENTIONS:
Drug: Ketamine Injectable Solution — 2 IM ketamine sessions with psychotherapy, spaced 9-15 days apart
  Arms: KAP (Ketamine-assisted Psychotherapy) Recipients
Other: Naturalistic Control — Continuation of pre-existing conventional treatment
  Arms: Naturalistic Comparator

SUMMARY:
The Conscious Dying/Conscious Living study will investigate the effect of KAP (ketamine-assisted psychotherapy) on individuals with terminal illness at five separate geographic locations. Two separate IM ketamine sessions will be administered to 18 subjects at each site, with psychotherapeutic support, including preparatory and integrative sessions. Assessments will be administered throughout the course of the protocol, which will take 4-6 weeks to complete, and the primary outcome measures are changes in the STAI (State-trait Anxiety Inventory, trait assessment only) and the DADDS (Death and Dying Distress Scale) from baseline at the beginning of the study to the conclusion of the treatment period. A six-subject naturalistic comparator group at each site will complete the same assessments without intervention, and then will be offered an optional crossover KAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Decision making capacity including conscious awareness and sufficient memory capacity.
* Ability to provide informed consent.
* Understanding of English language and ability to converse.
* 12 months or less life expectancy by prognosis.
* Age 18-85.
* Able to identify one or two Caregiver/Support Person(s) (relative, spouse, close friend, or other caregiver) who willing provide the following functions: 1) to drive the participant home on medication visits (if applicable), 2) to be reached by Clinical Investigator(s) in the event of a subject becoming suicidal or ill, and 3) to provide collateral information as needed. See Appendix D for Consent form.
* Have significant anxiety about impending death with a STAI Trait score of 45 or greater.
* If the individual has a documented history of anxiety disorder, the patient and investigator are in agreement that the individual's present anxiety is primarily resultant from or exacerbated by their illness and approaching death.
* May continue but not change psychiatric medications during the course of the study.
* May continue but not change therapists during the course of the study.
* Willing to refrain from using stimulants, anxiolytics, and PI designated medications during the day of the study sessions.
* Willing to refrain from using alcohol and marijuana for 24 hours before-- and the day of study sessions.
* Agrees to refrain from the use of any psychoactive drug during the course of the study., this referring to "Any drug that affects the nervous system leading to any or all of the following: Alterations in mood, awareness, thoughts, feelings, perception, cognition, or behavior.
* If necessary, are willing to be contacted via telephone on a daily basis by one of the therapists for a week after each experimental session

Exclusion Criteria:

* Clinical evidence of significant dementia or other cognitive impairment.
* Hypertension: Defined as Systolic greater than 145 or Diastolic greater than 95.
* History in intracranial bleeds or stroke.
* History of seizures.
* Known hypersensitivity to ketamine
* Class 2 or above heart disease.
* Below age 18 or above age 85.
* Subjects who are assessed to be at high risk of suicidal ideation or behavior.
* Have a history (or current diagnosis) of any of the following psychiatric disorders: a primary psychotic disorder, bipolar affective disorder type 1, dissociative identity disorder, an eating disorder (i.e., anorexia or bulimia), or a personality disorder that, in the opinion of the investigator, would interfere with the patient's participation in the study.
* IF receiving medication that may cause blunting of responses, and diminished affect such as antipsychotics, exclusion will be as per the evaluation of the PI and staff.
* Have evidence or history of significant (controlled or uncontrolled) cerebrovascular or cardiovascular disease, or any other medical disorder judged by the Principal Investigator(s) to significantly increase the risk of ketamine administration. Baseline Heart rate 110BPM or less; Greater than 50 BPM.
* Renal failure and dialysis.
* If on oxygen support, receiving no more than 4 liters
* Are experiencing cognitive and/or affective deficits as a result of ongoing chemotherapy that, in the opinion of the investigator, would interfere with the subject's ability to participate in the study.
* Have evidence or history of liver disease that would affect metabolism of ketamine. Transaminases do not exceed 3 times normal range
* Meet DSM-V criteria for substance abuse or dependence for any substance in the past sixty days except caffeine or nicotine-with the exception of opiates used prn for pain.
* Pregnant and Lactating Women
* Have any current problem, which in the opinion of the Principal Investigator(s) might interfere with participation in the study
* Are not able to give adequate informed consent
* Patients referred to our study who have by history electrolyte abnormalities (e.g., hypokalemia or hypomagnesemia), congestive heart failure, bradyarrhythmias, or patients taking concomitant medications that prolong the QT interval will be excluded as ondansetron may need to be used.
* Patients who are allergic to ondansetron will be excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) Form Y-2 (Trait Only) | 18-32 days
  Change in STAI (trait only) from baseline to conclusion of treatment (minimum 20/maximum 80, higher scores indicate increased anxiety and a worse outcome)
Death and Dying Distress Scale (DADDS) | 18-32 days
  Change in DADDS from baseline to conclusion of treatment (minimum 0/maximum 75, higher scores indicate increased death anxiety and a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Wolfson, MD, Principal Investigator — Ketamine Research Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrykowski MA, Cordova MJ, Studts JL, Miller TW. Posttraumatic stress disorder after treatment for breast cancer: prevalence of diagnosis and use of the PTSD Checklist-Civilian Version (PCL-C) as a screening instrument. J Consult Clin Psychol. 1998 Jun;66(3):586-90. doi: 10.1037//0022-006x.66.3.586. PMID 9642900
- [Background] Angrist B, d'Hollosy M, Sanfilipo M, Satriano J, Diamond G, Simberkoff M, Weinreb H. Central nervous system stimulants as symptomatic treatments for AIDS-related neuropsychiatric impairment. J Clin Psychopharmacol. 1992 Aug;12(4):268-72. PMID 1527230
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Barth J, Schumacher M, Herrmann-Lingen C. Depression as a risk factor for mortality in patients with coronary heart disease: a meta-analysis. Psychosom Med. 2004 Nov-Dec;66(6):802-13. doi: 10.1097/01.psy.0000146332.53619.b2. PMID 15564343
- [Background] Boston P, Bruce A, Schreiber R. Existential suffering in the palliative care setting: an integrated literature review. J Pain Symptom Manage. 2011 Mar;41(3):604-18. doi: 10.1016/j.jpainsymman.2010.05.010. Epub 2010 Dec 8. PMID 21145202
- [Background] Breitbart W, Rosenfeld B, Pessin H, Applebaum A, Kulikowski J, Lichtenthal WG. Meaning-centered group psychotherapy: an effective intervention for improving psychological well-being in patients with advanced cancer. J Clin Oncol. 2015 Mar 1;33(7):749-54. doi: 10.1200/JCO.2014.57.2198. Epub 2015 Feb 2. PMID 25646186
- [Background] Breen LJ, O'Connor M, Hewitt LY, Lobb EA. The "specter" of cancer: exploring secondary trauma for health professionals providing cancer support and counseling. Psychol Serv. 2014 Feb;11(1):60-7. doi: 10.1037/a0034451. Epub 2013 Sep 30. PMID 24079353
- [Background] Brown KW, Levy AR, Rosberger Z, Edgar L. Psychological distress and cancer survival: a follow-up 10 years after diagnosis. Psychosom Med. 2003 Jul-Aug;65(4):636-43. doi: 10.1097/01.psy.0000077503.96903.a6. PMID 12883115
- [Background] Bruera E, Driver L, Barnes EA, Willey J, Shen L, Palmer JL, Escalante C. Patient-controlled methylphenidate for the management of fatigue in patients with advanced cancer: a preliminary report. J Clin Oncol. 2003 Dec 1;21(23):4439-43. doi: 10.1200/JCO.2003.06.156. PMID 14645434
- [Background] Brundtland GH. From the World Health Organization. Mental health: new understanding, new hope. JAMA. 2001 Nov 21;286(19):2391. doi: 10.1001/jama.286.19.2391. No abstract available. PMID 11712923
- [Background] Busolo D, Woodgate R. Palliative care experiences of adult cancer patients from ethnocultural groups: a qualitative systematic review protocol. JBI Database System Rev Implement Rep. 2015 Jan;13(1):99-111. doi: 10.11124/jbisrir-2015-1809. PMID 26447011
- [Background] Carey LB, Hodgson TJ, Krikheli L, Soh RY, Armour AR, Singh TK, Impiombato CG. Moral Injury, Spiritual Care and the Role of Chaplains: An Exploratory Scoping Review of Literature and Resources. J Relig Health. 2016 Aug;55(4):1218-45. doi: 10.1007/s10943-016-0231-x. PMID 27094705
- [Background] Carney RM, Blumenthal JA, Catellier D, Freedland KE, Berkman LF, Watkins LL, Czajkowski SM, Hayano J, Jaffe AS. Depression as a risk factor for mortality after acute myocardial infarction. Am J Cardiol. 2003 Dec 1;92(11):1277-81. doi: 10.1016/j.amjcard.2003.08.007. PMID 14636903
- [Background] Carney RM, Freedland KE. Depression, mortality, and medical morbidity in patients with coronary heart disease. Biol Psychiatry. 2003 Aug 1;54(3):241-7. doi: 10.1016/s0006-3223(03)00111-2. PMID 12893100
- [Background] Carr DB, Goudas LC, Denman WT, Brookoff D, Staats PS, Brennen L, Green G, Albin R, Hamilton D, Rogers MC, Firestone L, Lavin PT, Mermelstein F. Safety and efficacy of intranasal ketamine for the treatment of breakthrough pain in patients with chronic pain: a randomized, double-blind, placebo-controlled, crossover study. Pain. 2004 Mar;108(1-2):17-27. doi: 10.1016/j.pain.2003.07.001. PMID 15109503
- [Background] Chang T, Glazko AJ. Biotransformation and disposition of ketamine. Int Anesthesiol Clin. 1974 Summer;12(2):157-77. doi: 10.1097/00004311-197412020-00018. No abstract available. PMID 4603048
- [Background] Chochinov HM, Hassard T, McClement S, Hack T, Kristjanson LJ, Harlos M, Sinclair S, Murray A. The patient dignity inventory: a novel way of measuring dignity-related distress in palliative care. J Pain Symptom Manage. 2008 Dec;36(6):559-71. doi: 10.1016/j.jpainsymman.2007.12.018. Epub 2008 Jun 24. PMID 18579340
- [Background] Clark JL, Kalan GE. Effective treatment of severe cancer pain of the head using low-dose ketamine in an opioid-tolerant patient. J Pain Symptom Manage. 1995 May;10(4):310-4. doi: 10.1016/0885-3924(95)00010-V. PMID 7541437
- [Background] Wolfson PE, Andries J, Feduccia AA, Jerome L, Wang JB, Williams E, Carlin SC, Sola E, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. MDMA-assisted psychotherapy for treatment of anxiety and other psychological distress related to life-threatening illnesses: a randomized pilot study. Sci Rep. 2020 Nov 24;10(1):20442. doi: 10.1038/s41598-020-75706-1. PMID 33235285
- [Background] Cordova MJ, Andrykowski MA, Kenady DE, McGrath PC, Sloan DA, Redd WH. Frequency and correlates of posttraumatic-stress-disorder-like symptoms after treatment for breast cancer. J Consult Clin Psychol. 1995 Dec;63(6):981-6. doi: 10.1037//0022-006x.63.6.981. PMID 8543720
- [Background] Dakwar E, Levin FR. The emerging role of meditation in addressing psychiatric illness, with a focus on substance use disorders. Harv Rev Psychiatry. 2009;17(4):254-67. doi: 10.1080/10673220903149135. PMID 19637074
- [Background] Dakwar E, Levin F, Foltin RW, Nunes EV, Hart CL. The effects of subanesthetic ketamine infusions on motivation to quit and cue-induced craving in cocaine-dependent research volunteers. Biol Psychiatry. 2014 Jul 1;76(1):40-6. doi: 10.1016/j.biopsych.2013.08.009. Epub 2013 Sep 12. PMID 24035344
- [Background] Dore J, Turnipseed B, Dwyer S, Turnipseed A, Andries J, Ascani G, Monnette C, Huidekoper A, Strauss N, Wolfson P. Ketamine Assisted Psychotherapy (KAP): Patient Demographics, Clinical Data and Outcomes in Three Large Practices Administering Ketamine with Psychotherapy. J Psychoactive Drugs. 2019 Apr-Jun;51(2):189-198. doi: 10.1080/02791072.2019.1587556. Epub 2019 Mar 27. PMID 30917760
- [Background] Feldman DB. Posttraumatic stress disorder at the end of life: extant research and proposed psychosocial treatment approach. Palliat Support Care. 2011 Dec;9(4):407-18. doi: 10.1017/S1478951511000435. PMID 22104417
- [Background] Fernandez F, Levy JK, Samley HR, Pirozzolo FJ, Lachar D, Crowley J, Adams S, Ross B, Ruiz P. Effects of methylphenidate in HIV-related depression: a comparative trial with desipramine. Int J Psychiatry Med. 1995;25(1):53-67. doi: 10.2190/16FH-9ECT-Y280-VV45. PMID 7649718
- [Background] Fernandez F, Adams F, Holmes VF, Levy JK, Neidhart M. Methylphenidate for depressive disorders in cancer patients. An alternative to standard antidepressants. Psychosomatics. 1987 Sep;28(9):455-61. doi: 10.1016/S0033-3182(87)72476-1. No abstract available. PMID 3432548
- [Background] Fine PG. Low-dose ketamine in the management of opioid nonresponsive terminal cancer pain. J Pain Symptom Manage. 1999 Apr;17(4):296-300. doi: 10.1016/s0885-3924(98)00144-4. PMID 10203883
- [Background] Fitzgibbon EJ, Hall P, Schroder C, Seely J, Viola R. Low dose ketamine as an analgesic adjuvant in difficult pain syndromes: a strategy for conversion from parenteral to oral ketamine. J Pain Symptom Manage. 2002 Feb;23(2):165-70. doi: 10.1016/s0885-3924(01)00393-1. PMID 11844639
- [Background] Fontana AE, Loschi JA. [Antidepressive therapy with C1 581]. Acta Psiquiatr Psicol Am Lat. 1974 Feb;20(1):32-9. No abstract available. Spanish. PMID 4455018
- [Background] Goldsmith RE, Gerhart JI, Chesney SA, Burns JW, Kleinman B, Hood MM. Mindfulness-based stress reduction for posttraumatic stress symptoms: building acceptance and decreasing shame. J Evid Based Complementary Altern Med. 2014 Oct;19(4):227-34. doi: 10.1177/2156587214533703. Epub 2014 May 7. PMID 24812075
- [Background] Grassi L, Costantini A. Psychosocial needs and well-being issues of long-term survivors and cured cancer patients. Epidemiol Prev. 2014 Nov-Dec;38(6 Suppl 1):126-9. No abstract available. English, Italian. PMID 25759297
- [Background] Grassi L, Caruso R, Hammelef K, Nanni MG, Riba M. Efficacy and safety of pharmacotherapy in cancer-related psychiatric disorders across the trajectory of cancer care: a review. Int Rev Psychiatry. 2014 Feb;26(1):44-62. doi: 10.3109/09540261.2013.842542. PMID 24716500
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Hardy SE. Methylphenidate for the treatment of depressive symptoms, including fatigue and apathy, in medically ill older adults and terminally ill adults. Am J Geriatr Pharmacother. 2009 Feb;7(1):34-59. doi: 10.1016/j.amjopharm.2009.02.006. PMID 19281939
- [Background] Hepgul N, King S, Amarasinghe M, Breen G, Grant N, Grey N, Hotopf M, Moran P, Pariante CM, Tylee A, Wingrove J, Young AH, Cleare AJ. Clinical characteristics of patients assessed within an Improving Access to Psychological Therapies (IAPT) service: results from a naturalistic cohort study (Predicting Outcome Following Psychological Therapy; PROMPT). BMC Psychiatry. 2016 Feb 27;16:52. doi: 10.1186/s12888-016-0736-6. PMID 26920578
- [Background] Hijazi Y, Boulieu R. Contribution of CYP3A4, CYP2B6, and CYP2C9 isoforms to N-demethylation of ketamine in human liver microsomes. Drug Metab Dispos. 2002 Jul;30(7):853-8. doi: 10.1124/dmd.30.7.853. PMID 12065445
- [Background] Homsi J, Nelson KA, Sarhill N, Rybicki L, LeGrand SB, Davis MP, Walsh D. A phase II study of methylphenidate for depression in advanced cancer. Am J Hosp Palliat Care. 2001 Nov-Dec;18(6):403-7. doi: 10.1177/104990910101800610. PMID 11712722
- [Background] Iglewicz A, Morrison K, Nelesen RA, Zhan T, Iglewicz B, Fairman N, Hirst JM, Irwin SA. Ketamine for the treatment of depression in patients receiving hospice care: a retrospective medical record review of thirty-one cases. Psychosomatics. 2015 Jul-Aug;56(4):329-37. doi: 10.1016/j.psym.2014.05.005. Epub 2014 Jun 5. PMID 25616995
- [Background] Iconomou G, Iconomou AV, Argyriou AA, Nikolopoulos A, Ifanti AA, Kalofonos HP. Emotional distress in cancer patients at the beginning of chemotherapy and its relation to quality of life. J BUON. 2008 Apr-Jun;13(2):217-22. PMID 18555468
- [Background] Irwin SA, Iglewicz A. Oral ketamine for the rapid treatment of depression and anxiety in patients receiving hospice care. J Palliat Med. 2010 Jul;13(7):903-8. doi: 10.1089/jpm.2010.9808. PMID 20636166
- [Background] Irwin SA, Iglewicz A, Nelesen RA, Lo JY, Carr CH, Romero SD, Lloyd LS. Daily oral ketamine for the treatment of depression and anxiety in patients receiving hospice care: a 28-day open-label proof-of-concept trial. J Palliat Med. 2013 Aug;16(8):958-65. doi: 10.1089/jpm.2012.0617. Epub 2013 Jun 27. PMID 23805864
- [Background] Jacobsen PB, Widows MR, Hann DM, Andrykowski MA, Kronish LE, Fields KK. Posttraumatic stress disorder symptoms after bone marrow transplantation for breast cancer. Psychosom Med. 1998 May-Jun;60(3):366-71. doi: 10.1097/00006842-199805000-00026. PMID 9625227
- [Background] Kannan TR, Saxena A, Bhatnagar S, Barry A. Oral ketamine as an adjuvant to oral morphine for neuropathic pain in cancer patients. J Pain Symptom Manage. 2002 Jan;23(1):60-5. doi: 10.1016/s0885-3924(01)00373-6. PMID 11779670
- [Background] Lapidus KA, Levitch CF, Perez AM, Brallier JW, Parides MK, Soleimani L, Feder A, Iosifescu DV, Charney DS, Murrough JW. A randomized controlled trial of intranasal ketamine in major depressive disorder. Biol Psychiatry. 2014 Dec 15;76(12):970-6. doi: 10.1016/j.biopsych.2014.03.026. Epub 2014 Apr 3. PMID 24821196
- [Background] Lara DR, Bisol LW, Munari LR. Antidepressant, mood stabilizing and procognitive effects of very low dose sublingual ketamine in refractory unipolar and bipolar depression. Int J Neuropsychopharmacol. 2013 Oct;16(9):2111-7. doi: 10.1017/S1461145713000485. Epub 2013 May 20. PMID 23683309
- [Background] Lauretti GR, Lima IC, Reis MP, Prado WA, Pereira NL. Oral ketamine and transdermal nitroglycerin as analgesic adjuvants to oral morphine therapy for cancer pain management. Anesthesiology. 1999 Jun;90(6):1528-33. doi: 10.1097/00000542-199906000-00005. PMID 10360847
- [Background] Lee H, Kim SW, Kim JM, Shin IS, Yang SJ, Yoon JS. Comparing effects of methylphenidate, sertraline and placebo on neuropsychiatric sequelae in patients with traumatic brain injury. Hum Psychopharmacol. 2005 Mar;20(2):97-104. doi: 10.1002/hup.668. PMID 15641125
- [Background] Little B, Chang T, Chucot L, Dill WA, Enrile LL, Glazko AJ, Jassani M, Kretchmer H, Sweet AY. Study of ketamine as an obstetric anesthetic agent. Am J Obstet Gynecol. 1972 May 15;113(2):247-60. doi: 10.1016/0002-9378(72)90774-0. No abstract available. PMID 4554554
- [Background] Lobb EA, Kristjanson LJ, Aoun SM, Monterosso L, Halkett GK, Davies A. Predictors of complicated grief: a systematic review of empirical studies. Death Stud. 2010 Sep;34(8):673-98. doi: 10.1080/07481187.2010.496686. PMID 24482845
- [Background] Lossignol DA, Obiols-Portis M, Body JJ. Successful use of ketamine for intractable cancer pain. Support Care Cancer. 2005 Mar;13(3):188-93. doi: 10.1007/s00520-004-0684-4. Epub 2004 Oct 6. PMID 15480820
- [Background] Luckenbaugh DA, Niciu MJ, Ionescu DF, Nolan NM, Richards EM, Brutsche NE, Guevara S, Zarate CA. Do the dissociative side effects of ketamine mediate its antidepressant effects? J Affect Disord. 2014 Apr;159:56-61. doi: 10.1016/j.jad.2014.02.017. Epub 2014 Feb 18. PMID 24679390
- [Background] Macleod AD. Methylphenidate in terminal depression. J Pain Symptom Manage. 1998 Sep;16(3):193-8. doi: 10.1016/s0885-3924(98)00071-2. PMID 9769622
- [Background] Manne SL, Du Hamel K, Gallelli K, Sorgen K, Redd WH. Posttraumatic stress disorder among mothers of pediatric cancer survivors: diagnosis, comorbidity, and utility of the PTSD checklist as a screening instrument. J Pediatr Psychol. 1998 Dec;23(6):357-66. doi: 10.1093/jpepsy/23.6.357. PMID 9824924
- [Background] Matsuo N, Morita T. Physician-reported practice of the use of methylphenidate in Japanese palliative care units. J Pain Symptom Manage. 2007 Jun;33(6):655-6. doi: 10.1016/j.jpainsymman.2007.02.025. No abstract available. PMID 17531905
- [Background] Mercadante S, Arcuri E, Ferrera P, Villari P, Mangione S. Alternative treatments of breakthrough pain in patients receiving spinal analgesics for cancer pain. J Pain Symptom Manage. 2005 Nov;30(5):485-91. doi: 10.1016/j.jpainsymman.2005.04.014. PMID 16310622
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Miyashita M, Morita T, Sato K, Hirai K, Shima Y, Uchitomi Y. Good death inventory: a measure for evaluating good death from the bereaved family member's perspective. J Pain Symptom Manage. 2008 May;35(5):486-98. doi: 10.1016/j.jpainsymman.2007.07.009. Epub 2008 Mar 20. PMID 18358685
- [Background] Patrick DL, Ferketich SL, Frame PS, Harris JJ, Hendricks CB, Levin B, Link MP, Lustig C, McLaughlin J, Reid LD, Turrisi AT 3rd, Unutzer J, Vernon SW; National Institutes of Health State-of-the-Science Panel. National Institutes of Health State-of-the-Science Conference Statement: Symptom management in cancer: pain, depression, and fatigue, July 15-17, 2002. J Natl Cancer Inst Monogr. 2004;(32):9-16. doi: 10.1093/jncimonographs/djg014. PMID 15263035
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Background] Satin JR, Linden W, Phillips MJ. Depression as a predictor of disease progression and mortality in cancer patients: a meta-analysis. Cancer. 2009 Nov 15;115(22):5349-61. doi: 10.1002/cncr.24561. PMID 19753617
- [Background] Schulz R, Monin JK, Czaja SJ, Lingler JH, Beach SR, Martire LM, Dodds A, Hebert RS, Zdaniuk B, Cook TB. Measuring the experience and perception of suffering. Gerontologist. 2010 Dec;50(6):774-84. doi: 10.1093/geront/gnq033. Epub 2010 May 17. PMID 20478899
- [Background] Stefanczyk-Sapieha L, Oneschuk D, Demas M. Intravenous ketamine "burst" for refractory depression in a patient with advanced cancer. J Palliat Med. 2008 Nov;11(9):1268-71. doi: 10.1089/jpm.2008.9828. PMID 19021495
- [Background] Subramaniam K, Subramaniam B, Steinbrook RA. Ketamine as adjuvant analgesic to opioids: a quantitative and qualitative systematic review. Anesth Analg. 2004 Aug;99(2):482-95, table of contents. doi: 10.1213/01.ANE.0000118109.12855.07. PMID 15271729
- [Background] Thase ME, Friedman ES, Biggs MM, Wisniewski SR, Trivedi MH, Luther JF, Fava M, Nierenberg AA, McGrath PJ, Warden D, Niederehe G, Hollon SD, Rush AJ. Cognitive therapy versus medication in augmentation and switch strategies as second-step treatments: a STAR*D report. Am J Psychiatry. 2007 May;164(5):739-52. doi: 10.1176/ajp.2007.164.5.739. PMID 17475733
- [Background] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Background] Ventegodt S, Morad M, Hyam E, Merrick J. Clinical holistic medicine: induction of spontaneous remission of cancer by recovery of the human character and the purpose of life (the life mission). ScientificWorldJournal. 2004 May 26;4:362-77. doi: 10.1100/tsw.2004.94. PMID 15175834
- [Background] Walker J, Sawhney A, Hansen CH, Ahmed S, Martin P, Symeonides S, Murray G, Sharpe M. Treatment of depression in adults with cancer: a systematic review of randomized controlled trials. Psychol Med. 2014 Apr;44(5):897-907. doi: 10.1017/S0033291713001372. Epub 2013 Jun 19. PMID 23778105
- [Background] Wallace AE, Kofoed LL, West AN. Double-blind, placebo-controlled trial of methylphenidate in older, depressed, medically ill patients. Am J Psychiatry. 1995 Jun;152(6):929-31. doi: 10.1176/ajp.152.6.929. PMID 7755127
- [Background] Wan LB, Levitch CF, Perez AM, Brallier JW, Iosifescu DV, Chang LC, Foulkes A, Mathew SJ, Charney DS, Murrough JW. Ketamine safety and tolerability in clinical trials for treatment-resistant depression. J Clin Psychiatry. 2015 Mar;76(3):247-52. doi: 10.4088/JCP.13m08852. PMID 25271445
- [Background] Weber F, Wulf H, Gruber M, Biallas R. S-ketamine and s-norketamine plasma concentrations after nasal and i.v. administration in anesthetized children. Paediatr Anaesth. 2004 Dec;14(12):983-8. doi: 10.1111/j.1460-9592.2004.01358.x. PMID 15601346
- [Background] Wieber J, Gugler R, Hengstmann JH, Dengler HJ. Pharmacokinetics of ketamine in man. Anaesthesist. 1975 Jun;24(6):260-3. PMID 1155748
- [Background] Wilson KG, Chochinov HM, Skirko MG, Allard P, Chary S, Gagnon PR, Macmillan K, De Luca M, O'Shea F, Kuhl D, Fainsinger RL, Clinch JJ. Depression and anxiety disorders in palliative cancer care. J Pain Symptom Manage. 2007 Feb;33(2):118-29. doi: 10.1016/j.jpainsymman.2006.07.016. PMID 17280918
- [Derived] Schipper S, Nigam K, Schmid Y, Piechotta V, Ljuslin M, Beaussant Y, Schwarzer G, Boehlke C. Psychedelic-assisted therapy for treating anxiety, depression, and existential distress in people with life-threatening diseases. Cochrane Database Syst Rev. 2024 Sep 12;9(9):CD015383. doi: 10.1002/14651858.CD015383.pub2. PMID 39260823
- See also: Use of the Classic Hallucinogen Psilocybin for Treatment of Existential Distress Associated with Cancer — https://link.springer.com/chapter/10.1007/978-1-4614-4866-2_17
- See also: Ketamine: Dreams and Realities — https://maps.org/images/pdf/books/K-DreamsKJansenMAPS.pdf